CLINICAL TRIAL: NCT02504541
Title: A 6-Month Safety Study of QuickShot™ Testosterone Administered Subcutaneously Once Each Week to Adult Males With Hypogonadism
Brief Title: Subcutaneous Testosterone Enanthate Safety in Adult Men Diagnosed With Hypogonadism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Antares Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QST-15-005
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Testosterone enanthate
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; testosterone enanthate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone enanthate auto-injector (Experimental): Testosterone enanthate 50 mg / 75 mg / 100 mg administered subcutaneously once each week with possible titration to a higher or lower dose at scheduled intervals during study.
  Interventions: Combination Product: Testosterone enanthate auto-injector

INTERVENTIONS:
Combination Product: Testosterone enanthate auto-injector — Dose Adjustment 50 mg or 75 mg or 100 mg based upon Testosterone levels
  Other Names: Testosterone; Testosterone enanthate; QuickShot® Testosterone (QST)

SUMMARY:
Evaluation of safety of a concentration controlled testosterone enanthate QuickShot Testosterone regimen administered subcutaneously once each week to adult males with hypogonadism.

DETAILED DESCRIPTION:
Safety assessments, including laboratory assessments, adverse events and injection site assessments, will be conducted for all patients at scheduled intervals during the Treatment Titration Period.

ELIGIBILITY:
Inclusion Criteria:

* Adult men ≥18 and ≤75 years of age with a documented history of hypogonadism
* Total testosterone levels < 300 ng/dL at two qualification visits
* Patients in good general health

Exclusion Criteria:

* Allergy to sesame or testosterone products
* BMI ≥ 40 kg/m2
* Hematocrit ≥ 52%
* History or current evidence of breast or prostate cancer
* Elevated prostate-specific antigen (PSA) for age.
* Abnormal digital rectal examination (DRE)
* Unstable psychiatric illnesses
* Obstructive uropathy of prostatic origin
* Poorly controlled diabetes
* Congestive heart failure
* Within 6 months of screening, myocardial infarction (MI), unstable angina leading to hospitalization, percutaneous coronary intervention, coronary artery bypass graft, uncontrolled cardiac arrhythmia, stroke transient ischemia attack, carotid revascularization, endovascular procedure, or surgical intervention for peripheral vascular disease.
* History or current treatment of thromboembolic disease.
* Use of adrenocorticotropic hormone (ACTH) or oral/depot corticosteroids within 6 weeks of screening.
* History of severe, untreated sleep apnea
* Subjects with any clinically significant medical condition which, in the opinion of the investigator, would make the subject an unsuitable candidate for enrollment in the study
* Positive serology for HIV, hepatitis B or hepatitis C
* Current evidence of drug or alcohol abuse.
* Skin conditions in injection site that could confound injection site assessments.
* Administration of other investigational compounds within one month of screening or 5 half-lives of the investigational compound, whichever is longer).
* Use of estrogen, gonadotropin-releasing hormone (GnRH) or growth hormone within 12 months of screening.
* Use of other androgens (DHEA), anabolic steroids, other sex hormones) or other substances/supplements know to affect the pharmacokinetics (PK) of testosterone enanthate
* Considered or scheduled surgical or dental procedures associated with blood loss ≥500 mL during study.
* Donation of plasma or blood within 56 days of screening or history of donation of > 50 mL of blood or plasma within 3 months of screening.
* Donation of plasma or blood during study

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Bedel, MD, Principal Investigator — Prestige Clinical Research
Locations (20):
- United States (20):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Tucson, Arizona
  - San Diego, California
  - Aventura, Florida
  - Brandon, Florida
  - Jacksonville, Florida
  - Shreveport, Louisiana
  - Elkridge, Maryland
  - Garden City, New York
  - New York, New York
  - Columbus, Ohio
  - Franklin, Ohio
  - Medford, Oregon
  - Charleston, South Carolina
  - Greer, South Carolina
  - Hurst, Texas
  - West Valley City, Utah
  - Olympia, Washington
  - Renton, Washington

REFERENCES:
- [Derived] Gittelman M, Jaffe JS, Kaminetsky JC. Safety of a New Subcutaneous Testosterone Enanthate Auto-Injector: Results of a 26-Week Study. J Sex Med. 2019 Nov;16(11):1741-1748. doi: 10.1016/j.jsxm.2019.08.013. Epub 2019 Sep 21. PMID 31551193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 133 patients were enrolled in this study. 113 (85.0%) patients completed the study (through the Follow-up Visit) and 20 (15.0%) patients prematurely withdrew from the study.
Pre-assignment Details: Although 21 sites participated in the study, only 19 sites enrolled patients in the United States. This study was intended to collect additional safety and exposure data, to ensure compliance and accuracy.
Period: Overall Study
Arm/Group | Testosterone Enanthate Auto-injector
Started | 133
Completed | 113
Not Completed | 20
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1
Not completed — Met Stopping Criteria | 1
Not completed — Protocol Violation | 2
Not completed — Termination by Sponsor | 1
Not completed — Other | 2
Not completed — Multiple | 5

BASELINE CHARACTERISTICS:
Population: Masked dose assignment based upon Testosterone levels; Individual patients may receive all three dose levels.
Arm/Group | Testosterone Enanthate Auto-injector
Number analyzed (Participants) | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 116
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 113
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 133

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events as a Measure of Safety of QuickShot™ Testosterone (QST) Administered Subcutaneously (SC) Once Each Week to Adult Males With Hypogonadism
Description: Number of participants experiencing adverse events that started on or after the first dose of QST, or existed prior to the first dose and woresened in severity or relatedness to QST after dosing, were evaluated in this population.
  Although a patient may have had 2 or more TEAEs or SAEs, the patient was counted only once within a SOC category. The same patient may have contributed to 2 or more preferred term categories. (Four patients had a total of 9 SAEs during the study)
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Testosterone Enanthate Auto-injector
Number analyzed (Participants) | 133
Participants
  Patients with any TEAE | 87
  Patients with any TEAE related to QST | 34
  Patients with SAE | 4
  Patients with TEAE leading to Discontinuation | 8
  Patients with QST related TEAE and discontinuation | 4

ADVERSE EVENTS:
Time Frame: 26 Weeks
Description: Treatment-emergent adverse events were defined as any event that started in the study on or after the first dosing of IP, or existed prior to the first dose and worsened in severity or relatedness to IP after dosing. Percentage was calculated using the number of patients in the column heading as the denominator.
Arm/Group | Testosterone Enanthate Auto-injector
All-Cause Mortality (participants affected / at risk) | 0/133
Serious Adverse Events (participants affected / at risk) | 4/133
Other Adverse Events (participants affected / at risk) | 68/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Enanthate Auto-injector (N=133)
Visual Impairment (Eye disorders) | 1 (1) — VISUAL CHANGES OF NON-NEUROLOGIC ETIOLOGY
APPENDICITIS (Infections and infestations) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
HYPOXIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1)
RIGHT KNEE SEPTIC ARTHRITIS (Infections and infestations) | 1 (1)
PRINZMETAL ANGINA (Cardiac disorders) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) — NON ST-SEGMENT ELEVATION MYOCARDIAL INFARCTION
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) — NON-SUSTAINED VENTRICULAR TACHYCARDIA
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Enanthate Auto-injector (N=133)
Upper respiratory tract infection (Infections and infestations) | 10 (10)
Nasopharyngitis (Infections and infestations) | 5 (5)
Urinary tract infection (Infections and infestations) | 4 (4)
Hematocrit increased (Investigations) | 11 (11)
Blood creatine phosphokinase increased (Investigations) | 5 (5)
PSA increased (Investigations) | 4 (4)
Injection site hemorrhage (General disorders) | 8 (8)
Injection site bruising (General disorders) | 5 (5)
Fatigue (General disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Prostatitis (Reproductive system and breast disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other